CLINICAL TRIAL: NCT06388044
Title: Acceptance and Commitment Therapy for Infertility Patients: A Case Series
Brief Title: ACT for Infertility: Case Series
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00115010
Record Dates: First submitted 2024-04-17; First posted 2024-04-29 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Infertility; Psychological Distress; Acceptance and Commitment Therapy; Psychological Flexibility
Keywords: Infertility; Psychological Flexibility; Acceptance and Commitment Therapy
MeSH Terms: conditions — Infertility | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acceptance and Commitment Therapy (Experimental): For those that enroll in the study, the therapist will see patients for 12 therapy sessions in the fertility clinic, with sessions lasting between 50 and 60 minutes. The therapist will offer both in-person and virtual sessions.
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Acceptance and Commitment Therapy (ACT) is a third-wave cognitive behavioral therapy. ACT aims to increase psychological flexibility through six core processes: acceptance, cognitive defusion, present-moment awareness, self as context, values, and committed action.

SUMMARY:
In the United States, around 19% of reproductive-aged couples suffer from infertility. The psychological distress associated with infertility is well-established; those diagnosed commonly experience depression and anxiety symptoms, diminished quality of life, and relationship dissatisfaction. In the current study, the investigators report on a case series, in which up to 10 infertility patients will receive 12 sessions of Acceptance and Commitment Therapy (ACT). The overarching goal for the current case series is to determine whether ACT might be well-suited for infertility patients experiencing distress. The specific aims are: 1) to describe the components of the intervention that was delivered; 2) to determine the extent to which infertility patients perceive a 12-session ACT intervention beneficial and acceptable; 3) to describe change in mood, stress, and ACT processes across 12 sessions of ACT; and 4) to highlight potential processes through which ACT might promote benefits to the patient by describing how change in mood, stress, and ACT processes relate to each other over the course of 12 sessions of ACT.

DETAILED DESCRIPTION:
In this study, the investigators present Acceptance and Commitment Therapy (ACT) as a potentially well-suited intervention for infertility patients, and they highlight mechanisms and processes through which ACT might benefit patients. They present a series of cases in which the therapist uses an ACT approach to treat individuals diagnosed with infertility.

The Duke University Health System includes a fertility clinic, which houses an embedded clinical psychology team. Patients at the fertility center can participate in individual psychotherapy and/ or group psychotherapy as part of their fertility treatment. An interventionist will provide psychotherapy to up to 10 individuals on the therapy waitlist. Patients will be eligible for the study if they: are at least 18 years old, have a diagnosis of infertility, speak English, and are not already participating in individual therapy. Patients will be excluded from the study if they endorse current suicidality and/ or self-harming behavior, current psychosis symptoms, and/ or current substance use.

For those that enroll in the study, patients will complete 12 therapy sessions in the fertility clinic, with sessions lasting between 50 and 60 minutes. Although sessions will vary across individuals, the therapist will aim to target the six core ACT processes in all cases. The therapist will offer both in-person and virtual sessions. Participants will complete a subset of questionnaires at each study session.

ELIGIBILITY:
Inclusion Criteria: Patients will be eligible if they

* are at least 18 years old
* have a diagnosis of infertility
* speak English
* are not already participating in individual therapy.

Exclusion Criteria: Patients will be excluded from the study if they

* endorse current suicidality and/ or self-harming behavior
* current psychosis symptoms
* and/ or current substance use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-06-26 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Acceptability of the Intervention | Week 6 (Session 6) and week 12 (Session 12).
  Patients will answer several questions about the extent to which they perceive the intervention to be beneficial and acceptable. Patients will answer questions using a 5-point Likert scale, with 1 being 'strongly disagree' and 5 being 'strongly agree.' The investigators will use this information descriptively--for each question, they will describe patient responses by identifying the percentage of patients that responded with each option (e.g., 7 out of 10 patients indicated that they strongly agreed with the following question: [question]).

SECONDARY OUTCOMES:
Change in Fertility Problem Inventory (FPI) | Week 1 (Session 1), week 6 (Session 6), and week 12 (session 12).
  The FPI is a 46-item self-report questionnaire that measures infertility-related stress. It includes a global stress score, as well as additional scores for four constructs: social concern, sexual concern, relationship concern, and need for parenthood. Patients will answer questions using a scale of 1 to 6, with higher scores reflecting greater distress.
Change in Patient Health Questionnaire 9 (PHQ-9) | PHQ-9: Week 1 (Session 1), week 6 (Session 6), and week 12 (session 12).
  The PHQ-9 is a 9-item self-report questionnaire that measures symptoms of depression. Participants answer questions using a scale of 0 to 3, with higher scores reflecting more and/ or more severe depression symptoms.
Change in Patient Health Questionnaire 2 (PHQ-2) | PHQ-2: Weeks 2 (Session 2), 3 (Session 3), 4 (Session 4), 5 (Session 5), 7 (Session 7), 8 (Session 8), 9 (Session 9), 10 (Session 10), and 11 (Session 11).
  The PHQ-2 is a 2-item self-report questionnaire that measures symptoms of depression. Participants answer questions using a scale of 0 to 3, with higher scores reflecting more and/ or more severe depression symptoms.
Change in Generalized Anxiety Disorder Questionnaire 7 (GAD-7) | GAD-7: Week 1 (Session 1), week 6 (Session 6), and week 12 (session 12).
  The GAD-7 is a 7-item self-report questionnaire that measures symptoms of generalized anxiety. Participants answer questions using a scale of 0 to 3, with higher scores reflecting more and/ or more severe anxiety symptoms.
Change in Generalized Anxiety Disorder Questionnaire 2 (GAD-2) | GAD-2: Weeks 2 (Session 2), 3 (Session 3), 4 (Session 4), 5 (Session 5), 7 (Session 7), 8 (Session 8), 9 (Session 9), 10 (Session 10), and 11 (Session 11).
  The GAD-2 is a 2-item self-report questionnaire that measures symptoms of generalized anxiety. Participants answer questions using a scale of 0 to 3, with higher scores reflecting more and/ or more severe anxiety symptoms.
Change in Modified Differential Emotions Scale (mDES) | Week 1 (Session 1), week 6 (Session 6), and week 12 (session 12).
  The mDES is a 20-item self-report questionnaire that measures the extent to which one has felt a range of emotions, including both negative and positive emotions. It includes a positive emotions score and a negative emotions score. Participants answer questions on a scale of 0 to 4, with higher scores reflecting more of that type of emotion.
Change in Comprehensive Assessment of Acceptance and Commitment Therapy (CompACT-15) | Week 1 (Session 1), week 3 (Session 3), week 6 (Session 6), week 9 (Session 9), and week 12 (Session 12).
  The CompACT-15 is a 15-item self-report questionnaire that measures several components of psychological flexibility, including openness to experience, behavioral awareness, and valued action. Patients will answer questions using a scale of 0 to 6, with higher scores reflecting greater levels of psychological flexibility.
Change in Intolerance of Uncertainty (IUS) | Week 1 (Session 1), week 3 (Session 3), week 6 (Session 6), week 9 (Session 9), and week 12 (Session 12).
  The IUS is a 27-item self-report questionnaire that measures emotional, cognitive, and behavioral reactions to uncertainty, the consequences of uncertainty, and attempts to control the future. Patients will answer questions using a scale of 1 to 5, with higher scores reflecting greater levels of intolerance.
Change in Valuing Questionnaire (VQ) | Week 1 (Session 1), week 3 (Session 3), week 6 (Session 6), week 9 (Session 9), and week 12 (Session 12).
  The VQ is a 10-item self-report questionnaire that measures the consistency with which an individual's behavior is aligned with his or her values. The VQ includes two constructs: progress and obstruction. Participants will answer questions using a scale of 0 to 6. On the progress subscale, higher scores reflect a greater level of consistency between one's values and behavior. On the obstruction subscale, higher scores reflect a greater level of inconsistency between one's values and behavior.
Change in Values-Based Behavior | All sessions, weeks 1-12.
  Measured by self-reported values of importance.

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda Merwin, PhD, Principal Investigator — Duke University
Locations (1):
- Duke North Pavilion, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bright K, Dube L, Hayden KA, Gordon JL. Effectiveness of psychological interventions on mental health, quality of life and relationship satisfaction for individuals and/or couples undergoing fertility treatment: a systematic review and meta-analysis protocol. BMJ Open. 2020 Jul 19;10(7):e036030. doi: 10.1136/bmjopen-2019-036030. PMID 32690514
- [Background] Cunha M, Galhardo A, Pinto-Gouveia J. Experiential avoidance, self-compassion, self-judgment and coping styles in infertility. Sex Reprod Healthc. 2016 Dec;10:41-47. doi: 10.1016/j.srhc.2016.04.001. Epub 2016 Apr 8. PMID 27938872
- [Background] Doyle, M., & Carballedo, A. (2014). Infertility and mental health. Advances in psychiatric treatment, 20(5), 297-303.
- [Background] Dube L, Bright K, Hayden KA, Gordon JL. Efficacy of psychological interventions for mental health and pregnancy rates among individuals with infertility: a systematic review and meta-analysis. Hum Reprod Update. 2023 Jan 5;29(1):71-94. doi: 10.1093/humupd/dmac034. PMID 36191078
- [Background] Dube L, Nkosi-Mafutha N, Balsom AA, Gordon JL. Infertility-related distress and clinical targets for psychotherapy: a qualitative study. BMJ Open. 2021 Nov 9;11(11):e050373. doi: 10.1136/bmjopen-2021-050373. PMID 34753757
- [Background] Hayes-Skelton, S. A., & Eustis, E. H. (2020). Experiential avoidance.
- [Background] Hayes, S. C., & Hofmann, S. G. (2018). Future directions in CBT and Evidence-based therapy. Process-based CBT: The science and core clinical competencies of cognitive behavioral therapy, 427-435.
- [Background] Peterson, B. D., & Eifert, G. H. (2011). Using acceptance and commitment therapy to treat infertility stress. Cognitive and Behavioral Practice, 18(4), 577-587.
- [Background] Schuette SA, Andrade FC, Woodward JT, Smoski MJ. Identifying modifiable factors associated with psychological health in women experiencing infertility. J Health Psychol. 2023 Oct;28(12):1143-1156. doi: 10.1177/13591053231185549. Epub 2023 Jul 4. PMID 37403402